CLINICAL TRIAL: NCT03056131
Title: Diacutaneous Fibrolysis, Effects on Tension Type Headache
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sara Cabanillas Barea (Other)
Responsible Party: Sponsor-Investigator, Sara Cabanillas Barea, PT, Universidad de Zaragoza
Organization: Universidad de Zaragoza (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PI15/0229
Record Dates: First submitted 2017-02-13; First posted 2017-02-17 (Actual); Last update posted 2018-05-02 (Actual); Status verified 2018-05

CONDITIONS: Tension-Type Headache
MeSH Terms: conditions — Tension-Type Headache

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Diacutaneous Fibrolysis Treatment (Experimental)
  Interventions: Device: Diacutaneous Fibrolysis
- Control Group (No Intervention)

INTERVENTIONS:
Device: Diacutaneous Fibrolysis — Diacutaneous Fibrolysis is a non invasive physiotherapeutic technique applied by means a set of metallic hooks having the advantage of allowing a deeper and more precise application, which could not be achieved manually
  Arms: Diacutaneous Fibrolysis Treatment

SUMMARY:
Tension Type Headache (TTH) is a frecuent type of headache disorder (about 1 person in 5 worldwide). Individuals with TTH typically present pericraneal tenderness and an increased cervical muscle tone.

The most common treatment in primary care consists mainly on analgesic medication. However, different techniques of manual therapy have been shown to be effective in the treatment of these patients. Diacutaneous fibrolysis shows clinical benefits in relieving symptoms of tension type headache, but there is no scientific evidence that analyzes this effects.

The hypothesis of this study was that adding treatment with diacutaneous fibrolysis to the usual conservative treatment has beneficial effects on different variables of the headache.

The aim of the study was to assess the effect of diacutaneous fibrolisis on intensity, frequency, duration of headache and cervical function in patients with tension type headache.

A randomized controlled clinical trial has been designed to evaluate the effectiveness of diacutaneous fibrolysis technique compared to usual general practicioner care in patientes with tension type headache.

The study protocol has been approved by the Clinical Research Ethics Committee from the Aragon Community and all patients provided written consent.

Eighty-two people with clinical diagnosis of TTH were randomized into a intervention group or a control group. Intervention group received three sessions of Diacutaneous Fibrolysis, while control group was advised to maintain their usual pharmacologic treatment. Pain intensity (VAS), frecuency, location, cervical range of motion, head forward position and pressure pain thresholds (PPTs) were measured at baseline, postintervention, and 1 month follow-up after treatment. The Spanish version of the HIT-6 Questionnaire was used to measure disability/function at baseline and follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Tension-Type Headache according to the criteria of ICDH-III.

Exclusion Criteria:

* Currently undergoing physiotherapy treatment for headache
* Modification of pharmacological treatment in the last month
* Presence of red flags

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2015-10; Primary Completion 2017-12 (Actual); Study Completion 2018-05 (Actual)

PRIMARY OUTCOMES:
Change in Pain Intensity | 10 days
  Visual Analog Scale (VAS)

SECONDARY OUTCOMES:
Change in Pain Frequency | 10 days
Pressure Pain Threshold | 10 days
  Pressure algometry
Pericraneal tenderness | 10 days
  Manual assessment
Cervical Range of motion | 10 days
  Cervical Range of Motion (CROM)
Dissability | 1 month
  HIT-6 Questionnaire

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cabanillas-Barea S, Perez-Guillen S, Lopez-de-Celis C, Rodriguez-Sanz J, Fanlo-Mazas P, Carrasco-Uribarren A. Effects of diacutaneous fibrolysis in patients with tension-type headache: A randomized controlled trial. PLoS One. 2023 Mar 27;18(3):e0273877. doi: 10.1371/journal.pone.0273877. eCollection 2023. PMID 36972231